CLINICAL TRIAL: NCT04886050
Title: A Phase 1, Open-Label, Randomized, Single-Dose Crossover Study to Evaluate the Bioavailability of an LC350189 Tablet Relative to an LC350189 Capsule in Healthy Subjects
Brief Title: Relative Bioavailability Study to Assess an LC350189 Tablet Compared to an LC350189 Capsule in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-GDCL007
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Gout; Hyperuricemia
Keywords: bioavailability; relative
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LC350189 Formulation A (Tablet) (Active Comparator): Each subject will be administered a single LC350189 200mg (QD) Tablet on Day 1 and Day 5, respectively.
  Interventions: Drug: LC350189 Tablet
- LC350189 Formulation B (Capsule) (Active Comparator): Each subject will be administered two LC350189 100mg (QD) Capsules (2 x 100-mg capsules) on Day 1 or Day 5, respectively.
  Interventions: Drug: LC350189 Capsule

INTERVENTIONS:
Drug: LC350189 Tablet — Subject will receive an LC350189 Tablet as single dose on Day 1 or Day 5
  Other Names: LC350189
  Arms: LC350189 Formulation A (Tablet)
Drug: LC350189 Capsule — Subject will receive an LC350189 Capsule as single dose on Day 1 or Day 5
  Other Names: LC350189
  Arms: LC350189 Formulation B (Capsule)

SUMMARY:
This is an open-label, randomized, crossover, single dose study. Two single doses of LC350189(tablet or capsule formulations) will be administered with a washout period of at least 4-day between the doses to investigate the relative bioavailability of LC350189 after administration via tablet formulation compared with capsule formulation and to evaluate basic systemic pharmacokinetic parameters of the tablet formulation compared to the capsule formulation of LC350189.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female 18 to 50 years of age, inclusive.
* The subject has a body mass index 18 to 32 kg/m2, inclusive, at screening.
* The subject is judged by the investigator to be in good general health, as determined by medical history, clinical laboratory assessments, vital sign measurements, 12 lead electrocardiogram (ECG) results, and physical examination findings at screening.
* The subject agrees to comply with all protocol requirements.
* The subject is able to provide written informed consent.

Exclusion Criteria:

* The subject has a medical history with any issues affecting absorption or metabolism, as judged by the investigator.
* The subject has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at screening.
* The subject has a positive test result for SARS-CoV-2 at screening.
* The subject has used any prescription (excluding hormonal birth control and hormone replacement therapy) or over the counter medications (except paracetamol [up to 2 g per day]), including herbal or nutritional supplements, within 14 days before the first dose of study drug or throughout the study.
* The subject has consumed grapefruit or grapefruit juice, Seville orange or Seville orange containing products (eg, marmalade), or caffeine- or xanthine containing products within 48 hours before the first dose of study drug or throughout the study.
* The subject is a smoker or has used nicotine or nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 6 months before the first dose of study drug.
* The subject has a history of alcohol abuse or drug addiction within the last year or excessive alcohol consumption (regular alcohol intake >21 units per week for male subjects and >14 units of alcohol per week for female subjects) (1 unit is equal to approximately ½ pint [200 mL] of beer, 1 small glass [100 mL] of wine, or 1 measure [25 mL] of spirits).
* The subject has a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at screening or before the first dose of study drug.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-07-31 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
The relative bioavailability of LC350189 after administration via tablet formulation compared with capsule formulation by assessment of the area under the plasma concentration-time curve from zero to infinity for the tablet formulation capsule formation | From baseline up to Day 8 (72 hours post on Day 5)
  Blood sample for determination of plasma concentration of LC350189 will be collected at pre-dose and 0.5,1,2,4,6,8,16,24,36,48, and 72 hours

SECONDARY OUTCOMES:
Incidence of Adverse events | From baseline up to Day 8
  Safety assessment

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be determined